CLINICAL TRIAL: NCT02874391
Title: Use of Arterio-venous Fistula as First Choice for Intravenous Drug Administration in Kidney Transplant Recipients
Acronym: PerFAV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHRIP-15-633
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Evaluate the Risks of Using Arteriovenous Fistula as First Choise for Drug Administration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- AV fistula group
- Control group

SUMMARY:
Use of arteriovenous fistula for IV drug administration is controversial and often prohibited by nephrologists. However, we have been using this method in our department for years now in order to keep the patients 'veins for other fistulas in the future. The aim of this study is to evaluate our practice and maybe provide a justification for a larger multi-center study given the importance of this subject in patients with chronic renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years, functional AV fistula, new kidney transplant recipient

Exclusion Criteria:

* Prothetic AV fistula, Very recent AV fistula of less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the risk of complications of AV fistula | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Roux, Principal Investigator — University Hospital, Angers
Locations (1):
- CHU Angers, Angers, France